CLINICAL TRIAL: NCT00796601
Title: A 6-month, Double-blind, Placebo-controlled, Multi-center, Parallel Group, Maintenance Of Effect Study Of Esreboxetine (Pnu-165442g) Administered Once Daily (qd) In Patients With Fibromyalgia
Brief Title: Maintenance of Efficacy.
Status: Withdrawn | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: A6061054; A6061054; 2008-006760-10 (EudraCT Number)
Record Dates: First submitted 2008-11-20; First posted 2008-11-24 (Estimated); Last update posted 2018-11-29 (Actual); Status verified 2018-11

CONDITIONS: Fibromyalgia
Keywords: double-blind placebo-controlled maintenance of efficacy
MeSH Terms: conditions — Fibromyalgia | interventions — esreboxetine

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Esreboxetine (Experimental)
  Interventions: Drug: Esreboxetine
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Esreboxetine — Film coated tablets (2, 6, 8, 10 mg esreboxetine), once daily for 6 months
  Arms: Esreboxetine
Drug: Placebo — Film coated tablets (0 mg esreboxetine), once daily for 6 months
  Arms: Placebo

SUMMARY:
The hypothesis of Study A6061054 is to demonstrate superiority of efficacy of esreboxetine at 3 and 6 months compared to placebo.

ELIGIBILITY:
Inclusion Criteria:

* Subjects must meet the American College of Rheumatology (ACR) criteria for fibromyalgia
* Pain score greater than or equal to 4 on an 11-point NRS
* FIQ-Total score greater than or equal to 45 points

Exclusion Criteria:

* Other severe pain that may confound assessment or self evaluation of the pain associated with fibromyalgia
* Any autoimmune rheumatic disorder, non-focal rheumatic disease (other than fibromyalgia), clinically significant active infection, or untreated endocrine disorder
* Uncontrolled hypertension Pending Worker's Compensation; Current or recent diagnosis or episode of major depressive disorder, dysthymia and/or uncontrolled depression; Subjects to be at risk of suicide;

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-05-01 (Actual); Primary Completion 2010-05-01 (Estimated); Study Completion 2010-11-01 (Estimated)

PRIMARY OUTCOMES:
Change from baseline to 3 and 6 months in the mean daily pain rating score measured by the 11 point pain intensity Numerical Rating Scale (NRS). | 6 months
Change from baseline to 3 and 6 months in the FIQ-Total score | 6 months

SECONDARY OUTCOMES:
Pain (including other measures of daily pain and responder analyses); | 6 months
Function (including sub-scales of the FIQ, responder analyses of FIQ and SF-36); | 6 months
Global efficacy measures PGIC); | 6 months
Sleep (MOS); | 6 months
Work productivity; | 6 months
Depression (HADS) | 6 months
Safety (vital signs, ECG, laboratory, suicidal ideation) | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer

IPD SHARING:
Plan to Share IPD: Yes
Information relating to our policy on data sharing and the process for requesting data can be found at the following link: http://www.pfizer.com/research/clinical_trials/trial_data_and_results/data_requests

REFERENCES:
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A6061054&StudyName=Maintenance%20of%20efficacy.